CLINICAL TRIAL: NCT00626275
Title: A Phase 2a Randomized, Placebo- and Active-Controlled, Single-Dose, 3-Period, Crossover Study Followed by a Randomized, Placebo-Controlled, 14-Day, Parallel-Group Study Evaluating the Analgesic Efficacy and Safety of ADL5859 in Subjects With Rheumatoid Arthritis
Brief Title: Study Evaluating the Analgesic Efficacy and Safety of ADL5859 in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33CL232
Record Dates: First submitted 2008-02-22; First posted 2008-02-29 (Estimated); Results first posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — N,N-diethyl-4-(5-hydroxyspiro(chromene-2,4'-piperidine)-4-yl)benzamide; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ADL5859 -- 200 mg (Part A) (Experimental): ADL5859: 200 milligrams (mg), capsules, administered orally as a single dose during 1 of 3 Treatment Periods in Part A of the study
  Interventions: Drug: ADL5859
- Naproxen -- 500 mg (Part A) (Active Comparator): Naproxen: 500 mg, capsules, administered orally as a single dose during 1 of 3 Treatment Periods in Part A of the study
  Interventions: Drug: Naproxen
- Placebo (Part A) (Placebo Comparator): Matching placebo, capsules, administered orally, as a single dose during 1 of 3 Treatment Periods in Part A of the study
  Interventions: Drug: Placebo
- ADL5859 - 100 mg (Part B) (Experimental): ADL5859: 100 mg, capsules, administered orally, twice daily (BID) for 2 weeks during Part B of the study
  Interventions: Drug: ADL5859
- Placebo (Part B) (Placebo Comparator): Matching placebo, capsules, administered orally, BID for 2 weeks during Part B of the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADL5859
  Other Names: ADL-5859
  Arms: ADL5859 -- 200 mg (Part A)
Drug: Naproxen
  Other Names: Naprosyn
  Arms: Naproxen -- 500 mg (Part A)
Drug: Placebo
  Other Names: Lactose Monohydrate National Formulary (NF)
  Arms: Placebo (Part A)
Drug: ADL5859
  Other Names: ADL-5859
  Arms: ADL5859 - 100 mg (Part B)
Drug: Placebo
  Other Names: Lactose Monohydrate NF
  Arms: Placebo (Part B)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of ADL5859 in relieving pain associated with rheumatoid arthritis (RA) compared with placebo and naproxen (similar to Aleve®). A second objective is to see whether the effect of ADL5859 differs after a single dose compared with multiple doses.

DETAILED DESCRIPTION:
This Phase 2a study was conducted in 2 parts. Part A was a randomized, single-dose, double-blind, placebo- and active-controlled, 3-way crossover phase during which participants were administered study medication in the clinical facility. Part B was a 14-day, randomized, double-blind, placebo-controlled, parallel-group, multiple-dose phase in which participants self-administered study medication at home.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 18 and 75 years of age, inclusive
* Have a documented history of rheumatoid arthritis (diagnosed according to American College of Rheumatology criteria)
* Have painful rheumatoid arthritis with pain predominantly in the lower extremities (that is, hip, knees, ankles, and/or feet)
* Have an evoked lower extremity pain intensity (ELEPI) score of 5 or higher on a numeric pain rating scale (NPRS) completed on Day 1 of Part A before dosing (after resting for 45 minutes and then walking for at least 10 minutes on a treadmill) and then have a minimum ELEPI score of 4 on other visits during Part A
* If receiving disease modifying antirheumatic drugs, have a stable dose regimen for at least 30 days before study entry (90 days before study entry for biologic therapy)
* If biologic therapy has been recently discontinued, Enbrel™ or Orencia™ must have been discontinued at least 30 days before study entry, and Humira™, Remicade™, and Rituxan™ must have been discontinued at least 60 days before study entry
* For male participants, be surgically sterile or agree to use an appropriate method of contraception
* For female participants of child bearing potential, be surgically sterile or using an insertable, injectable, transdermal, or combination oral contraceptive deemed highly effective by the US Food and Drug Administration (FDA) through the completion of the study and have negative findings on a urine pregnancy test before administration of study medication (women who are postmenopausal [no menses for at least 2 years] are also eligible to participate)
* Have a body weight of at least 45 kilograms (kg)
* Be able to understand and comply with the protocol requirements (such as repeated treadmill walking and diary completion via the interactive voice response system), instructions, and protocol-specified restrictions.

Exclusion Criteria:

* Have an overall pain intensity (OPI) score equal to 10 at screening or before the first dose of study medication in Part A
* Have a pain intensity score for the upper body (that is, back, neck, fingers, wrists, elbows, and/or shoulders) above 7 on a numeric pain rating scale (NPRS) before study medication administration
* Have a history of headache requiring prescription treatment within 6 months of study entry
* Have significant renal disease (as indicated by blood urea nitrogen or serum creatinine ≥ 2 times the upper limit of normal) or have significant hepatic disease (as indicated by liver function test results ≥ 2 times the upper limit of normal)
* Have evidence of symptomatic orthostatic hypotension
* Have a history of a seizure disorder, including febrile seizures
* Have, as determined by the investigator or the sponsor's medical monitor, a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other conditions that would affect study participation
* Are taking cytochrome P450 (CYP) 3A4/5 or P glycoprotein (P gp) transporter inhibitors
* Have taken oral steroids within 30 days of study entry or intra articular steroids within 60 days of study entry (inhaled or topical steroids or stable oral dose ≤ 10 mg is permitted)
* Have a history or presence of allergy or intolerance to nonsteroidal anti-inflammatory drugs or acetaminophen, or have a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the study
* Have a history of alcoholism or drug addiction or abuse within 5 years before the scheduled administration of study medication
* Have participated in a trial of any investigational medication within 30 days before study drug administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Berger, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (8):
- United States (8):
  - New England Research Associates, Trumbull, Connecticut
  - Covance Clinical Research Unit Inc., Daytona Beach, Florida
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Winthrop University Hospital, Clinical Trials Center, Mineola, New York
  - University Hospitals Case Medical Center, Division of Rheumatology, Rheumatology Clinical Research Unit, Beachwood, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A, Sequence 1: Placebo First, Then ADL5859, Then Naproxen: Eligible participants were randomized to 1 of 6 treatment sequences. Each treatment sequence had 3 treatment periods, each separated by a washout period of at least 48 hours and up to 1 week between doses. During each treatment period of Part A, participants received a single dose of study medication (placebo, then ADL5859 200 milligrams (mg), then naproxen 500 mg).
  Part A, Treatment Period 1: matching placebo, capsules, administered orally, as a single dose; Part A, Treatment Period 2: ADL5859 200 mg, capsules, administered orally as a single dose; and Part A, Treatment Period 3: naproxen 500 mg, capsules, administered orally as a single dose
- Part A Sequence 2: ADL5859 First, Then Naproxen, Then Placebo: Eligible participants were randomized to 1 of 6 treatment sequences. Each treatment sequence had 3 treatment periods, each separated by a washout period of at least 48 hours and up to 1 week between doses. During each treatment period of Part A, participants received a single dose of study medication (ADL5859 200 mg, then naproxen 500 mg, then placebo).
  Part A, Treatment Period 1: ADL5859 200 mg, capsules, administered orally as a single dose; Part A, Treatment Period 2: naproxen 500 mg, capsules, administered orally as a single dose; and Part A, Treatment Period 3: matching placebo, capsules, administered orally, as a single dose.
- Part A Sequence 3: Naproxen First, Then Placebo, Then ADL5859: Eligible participants were randomized to 1 of 6 treatment sequences. Each treatment sequence had 3 treatment periods, each separated by a washout period of at least 48 hours and up to 1 week between doses. During each treatment period of Part A, participants received a single dose of study medication (naproxen 500 mg, then placebo, then ADL5859 200 mg).
  Part A, Treatment Period 1: naproxen 500 mg, capsules, administered orally as a single dose; Part A, Treatment Period 2: matching placebo, capsules, administered orally, as a single dose; and Part A, Treatment Period 3: ADL5859 200 mg, capsules, administered orally as a single dose.
- Part A Sequence 4: Naproxen First, Then ADL5859, Then Placebo: Eligible participants were randomized to 1 of 6 treatment sequences. Each treatment sequence had 3 treatment periods, each separated by a washout period of at least 48 hours and up to 1 week between doses. During each treatment period of Part A, participants received a single dose of study medication (naproxen 500 mg, then ADL5859 200 mg, then placebo).
  Part A, Treatment Period 1: naproxen 500 mg, capsules, administered orally as a single dose; Part A, Treatment Period 2: ADL5859 200 mg, capsules, administered orally as a single dose; and Part A, Treatment Period 3: matching placebo, capsules, administered orally, as a single dose.
- Part A Sequence 5: Placebo First, Then Naproxen, Then ADL5859: Eligible participants were randomized to 1 of 6 treatment sequences. Each treatment sequence had 3 treatment periods, each separated by a washout period of at least 48 hours and up to 1 week between doses. During each treatment period of Part A, participants received a single dose of study medication (placebo, then naproxen 500 mg, then ADL5859 200 mg).
  Part A, Treatment Period 1: matching placebo, capsules, administered orally, as a single dose; Part A, Treatment Period 2: naproxen 500 mg, capsules, administered orally as a single dose; and Part A, Treatment Period 3: ADL5859 200 mg, capsules, administered orally as a single dose.
- Part A Sequence 6: ADL5859 First, Then Placebo, Then Naproxen: Eligible participants were randomized to 1 of 6 treatment sequences. Each treatment sequence had 3 treatment periods, each separated by a washout period of at least 48 hours. During each treatment period of Part A, participants received a single dose of study medication (ADL5859 200 mg, then placebo, then naproxen 500 mg).
  Part A, Treatment Period 1: ADL5859 200 mg, capsules, administered orally as a single dose; Part A, Treatment Period 2: matching placebo, capsules, administered orally, as a single dose; and Part A, Treatment Period 3: naproxen 500 mg, capsules, administered orally as a single dose.
- Part B: ADL5859 100 mg: ADL5859: 100 mg, capsules, administered orally, twice daily (BID) for 2 weeks during Part B of the study
- Part B: Placebo: Matching placebo, capsules, administered orally, BID for 2 weeks during Part B of the study
Period: Part A - Treatment Period 1
Arm/Group | Part A, Sequence 1: Placebo First, Then ADL5859, Then Naproxen | Part A Sequence 2: ADL5859 First, Then Naproxen, Then Placebo | Part A Sequence 3: Naproxen First, Then Placebo, Then ADL5859 | Part A Sequence 4: Naproxen First, Then ADL5859, Then Placebo | Part A Sequence 5: Placebo First, Then Naproxen, Then ADL5859 | Part A Sequence 6: ADL5859 First, Then Placebo, Then Naproxen | Part B: ADL5859 100 mg | Part B: Placebo
Started | 7 | 7 | 7 | 8 | 9 | 8 | 0 | 0
Received at Least 1 Dose of Study Drug | 7 | 7 | 7 | 8 | 9 | 8 | 0 | 0
Completed | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part A - Washout Period 1
Arm/Group | Part A, Sequence 1: Placebo First, Then ADL5859, Then Naproxen | Part A Sequence 2: ADL5859 First, Then Naproxen, Then Placebo | Part A Sequence 3: Naproxen First, Then Placebo, Then ADL5859 | Part A Sequence 4: Naproxen First, Then ADL5859, Then Placebo | Part A Sequence 5: Placebo First, Then Naproxen, Then ADL5859 | Part A Sequence 6: ADL5859 First, Then Placebo, Then Naproxen | Part B: ADL5859 100 mg | Part B: Placebo
Started | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Completed | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A - Treatment Period 2
Arm/Group | Part A, Sequence 1: Placebo First, Then ADL5859, Then Naproxen | Part A Sequence 2: ADL5859 First, Then Naproxen, Then Placebo | Part A Sequence 3: Naproxen First, Then Placebo, Then ADL5859 | Part A Sequence 4: Naproxen First, Then ADL5859, Then Placebo | Part A Sequence 5: Placebo First, Then Naproxen, Then ADL5859 | Part A Sequence 6: ADL5859 First, Then Placebo, Then Naproxen | Part B: ADL5859 100 mg | Part B: Placebo
Started | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Received at Least 1 Dose of Study Drug | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Completed | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A - Washout Period 2
Arm/Group | Part A, Sequence 1: Placebo First, Then ADL5859, Then Naproxen | Part A Sequence 2: ADL5859 First, Then Naproxen, Then Placebo | Part A Sequence 3: Naproxen First, Then Placebo, Then ADL5859 | Part A Sequence 4: Naproxen First, Then ADL5859, Then Placebo | Part A Sequence 5: Placebo First, Then Naproxen, Then ADL5859 | Part A Sequence 6: ADL5859 First, Then Placebo, Then Naproxen | Part B: ADL5859 100 mg | Part B: Placebo
Started | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Completed | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A - Treatment Period 3
Arm/Group | Part A, Sequence 1: Placebo First, Then ADL5859, Then Naproxen | Part A Sequence 2: ADL5859 First, Then Naproxen, Then Placebo | Part A Sequence 3: Naproxen First, Then Placebo, Then ADL5859 | Part A Sequence 4: Naproxen First, Then ADL5859, Then Placebo | Part A Sequence 5: Placebo First, Then Naproxen, Then ADL5859 | Part A Sequence 6: ADL5859 First, Then Placebo, Then Naproxen | Part B: ADL5859 100 mg | Part B: Placebo
Started | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Received at Least 1 Dose of Study Drug | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Completed | 6 | 7 | 6 | 8 | 9 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Re-randomization Period for Part B
Arm/Group | Part A, Sequence 1: Placebo First, Then ADL5859, Then Naproxen | Part A Sequence 2: ADL5859 First, Then Naproxen, Then Placebo | Part A Sequence 3: Naproxen First, Then Placebo, Then ADL5859 | Part A Sequence 4: Naproxen First, Then ADL5859, Then Placebo | Part A Sequence 5: Placebo First, Then Naproxen, Then ADL5859 | Part A Sequence 6: ADL5859 First, Then Placebo, Then Naproxen | Part B: ADL5859 100 mg | Part B: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 24
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 24
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A, Sequence 1: Placebo First, Then ADL5859, Then Naproxen | Part A Sequence 2: ADL5859 First, Then Naproxen, Then Placebo | Part A Sequence 3: Naproxen First, Then Placebo, Then ADL5859 | Part A Sequence 4: Naproxen First, Then ADL5859, Then Placebo | Part A Sequence 5: Placebo First, Then Naproxen, Then ADL5859 | Part A Sequence 6: ADL5859 First, Then Placebo, Then Naproxen | Part B: ADL5859 100 mg | Part B: Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 24
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 23
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- All Treated Participants: All participants who received at least 1 dose of study drug during any sequence of Part A of the study. Baseline measures reported in aggregate for all participants to avoid double counting of Parts A and B.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Part A: Average Difference Between Baseline and Post Dose Evoked (by Treadmill Walking) Lower-Extremity Pain Intensity Scores (AELEPID) Over the 6 Hours After Dosing
Description: Approximately 1 hour before baseline and again approximately 45 minutes before the 2-, 4-, and 6-hour time points, participants rested for 45 minutes, then they started the treadmill walk at 15 minutes before baseline and at the 2-, 4-, and 6-hour time points. After the treadmill walk, participants were asked to rate their lower extremity pain on an 11 point Numeric Pain Rating Scale (NPRS), with 0 indicating No Pain and 10 indicating Worst Possible Pain. The average difference between baseline and 6 hours post dose evoked lower-extremity pain intensity scores (AELEPID-6) is presented for each treatment group. Difference = predose (baseline) NPRS score - NPRS score 6 hours post dose.
  Least square (LS) means and standard errors (SE) were calculated from an analysis-of-covariance (ANCOVA) model with fixed effects for sequence, treatment, period, predose evoked lower extremity pain intensity as a covariate, and a random effect for participant nested within sequence.
Time Frame: Baseline through 6 hours post dose
Population: Participants in Part A who received at least 1 dose of study drug and had at least 1 pain intensity assessment post dose.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Naproxen - 500 mg (Part A): Naproxen: 500 mg, capsules, administered orally as a single dose during 1 of 3 Treatment Periods in Part A of the study
- ADL5859 - 200 mg (Part A): ADL5859: 200 mg, capsules, administered orally as a single dose during 1 of 3 Treatment Periods in Part A of the study
Arm/Group | Placebo (Part A) | Naproxen - 500 mg (Part A) | ADL5859 - 200 mg (Part A)
Number analyzed (Participants) | 45 | 45 | 44
units on a scale | 1.12 (0.240) | 1.95 (0.240) | 1.20 (0.242)

2. Secondary Outcome: Part A: Pain Intensity Score (NPRS Score) for Overall Pain, for Lower Extremity Pain, and for Evoked (by Treadmill Walking) Lower Extremity Pain
Description: Overall Pain Intensity (OPI), "Now" Lower Extremity Pain Intensity (LEPI), and Evoked Lower Extremity Pain Intensity (ELEPI) were assessed using the 11-point Numeric Pain Rating Scale (NPRS), with 0 indicating No Pain and 10 indicating Worst Possible Pain. OPI was assessed at 15 minutes before dosing for baseline and at 6 and 12 hours (hr) after dosing. At 15 minutes before dosing, during Period 1 only, participants were also asked to assess their average LEPI over the last 24 hours as a baseline measurement. "Now" LEPI was assessed at 15 minutes before dosing for baseline and at the 1-, 2-, 3-, 4-, 5-, 6-, and 12-hour time points. Approximately 1 hour before dosing and approximately 45 minutes before the 2-, 4-, and 6-hour time points, the participant rested for 45 minutes, then (after the "Now" LEPI assessment) he or she started a treadmill walk at 15 minutes before dosing for baseline and at the 2-, 4-, and 6-hour time points, and then assessed ELEPI.
Time Frame: Baseline up to 12 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Part A) | Naproxen - 500 mg (Part A) | ADL5859 - 200 mg (Part A)
Number analyzed (Participants) | 45 | 45 | 44
units on a scale
  ELEPI, Baseline | 6.36 (1.873) | 6.20 (1.471) | 6.363 (1.806)
  ELEPI, 2 hr Post Dose | 5.47 (1.854) | 4.71 (1.973) | 5.45 (1.649)
  ELEPI, 4 hr Post Dose | 5.16 (2.174) | 4.24 (1.760) | 5.00 (2.035)
  ELEPI, 6 hr Post Dose | 4.93 (2.517) | 4.00 (1.871) | 4.95 (2.124)
  LEPI, Baseline | 6.18 (2.059) | 5.78 (1.845) | 5.68 (1.840)
  LEPI, 1 hr Post Dose | 5.38 (2.124) | 5.00 (1.719) | 5.34 (1.584)
  LEPI, 2 hr Post Dose | 5.24 (2.013) | 4.33 (1.822) | 4.91 (1.507)
  LEPI, 3 hr Post Dose | 4.67 (2.089) | 4.04 (1.858) | 4.73 (1.590)
  LEPI, 4 hr Post Dose | 4.76 (2.036) | 3.93 (1.737) | 4.70 (1.593)
  LEPI, 5 hr Post Dose | 4.71 (2.117) | 3.98 (1.685) | 4.73 (1.921)
  LEPI, 6 hr Post Dose | 4.49 (2.149) | 3.89 (1.774) | 4.77 (1.696)
  LEPI, 12 hr Post Dose | 5.11 (2.037) | 3.78 (1.813) | 4.76 (1.817)
  OPI, Baseline | 6.20 (1.89) | 6.13 (1.753) | 5.77 (1.710)
  OPI, 6 hr Post Dose | 4.80 (2.282) | 4.04 (1.833) | 4.91 (1.815)
  OPI, 12 hr Post Dose | 5.03 (1.993) | 3.73 (1.880) | 4.89 (1.955)

3. Secondary Outcome: Part B: Mean Daily LEPI Scores for Weeks 1 and 2
Description: Participants assessed their "Now" LEPI 3 times each day (morning, midday, and evening at approximately 10 AM, 2 PM, and 8 PM) and before taking any rescue medication. At each time point, participants were asked to rate their lower extremity pain on an 11 point Numeric Pain Rating Scale (NPRS), with 0 indicating No Pain and 10 indicating Worst Possible Pain. If a scheduled pain assessment was taken within 4 hours of rescue medication, the observed pain score was replaced by the pain score obtained right before the rescue medication was taken.
Time Frame: Baseline through Week 1 and Week 1 through Week 2
Population: Participants in Part B who received at least 1 dose of study drug and had at least 1 pain intensity assessment post dose.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ADL5859 - 100 mg (Part B): ADL5859: 100 mg, capsules, administered orally, BID for 2 weeks during Part B of the study
Arm/Group | Placebo (Part B) | ADL5859 - 100 mg (Part B)
Number analyzed (Participants) | 24 | 20
units on a scale
  Over Week 1 | 4.28 (1.691) | 4.17 (1.667)
  Over Week 2 | 4.23 (2.090) | 4.13 (1.756)

4. Secondary Outcome: Part A: Pain Intensity Difference Between Baseline and the Value at Each Scheduled Time Point for Overall Pain
Description: Overall Pain Intensity (OPI) was assessed by the participant using the 11-point Numeric Pain Rating Scale (NPRS), with 0 indicating No Pain and 10 indicating Worst Possible Pain. OPI was assessed at 15 minutes before dosing for baseline and at 6 and 12 hours after dosing. Difference = predose (baseline) OPI score - OPI score 6 and 12 hours post dose.
Time Frame: Baseline, 6 and 12 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo (Part A): Matching placebo capsules, administered orally, as a single dose during 1 of 3 Treatment Periods in Part A of the study
- ADL5859 - 200mg (Part A): ADL5859: 200 mg, capsules, administered orally as a single dose during 1 of 3 Treatment Periods in Part A of the study
Arm/Group | Placebo (Part A) | Naproxen - 500 mg (Part A) | ADL5859 - 200mg (Part A)
Number analyzed (Participants) | 45 | 45 | 44
units on a scale
  Change From Baseline 6 Hours Post Dose | 1.40 (2.240) | 2.09 (1.917) | 0.86 (2.120)
  Change From Baseline 12 Hours Post Dose | 1.16 (1.911) | 3.73 (1.880) | 0.92 (2.278)

5. Secondary Outcome: Part A: Average Difference Between Baseline and Postdose Evoked Lower Extremity Pain Over the 4 Hours After Dosing
Description: Evoked Lower Extremity Pain Intensity (ELEPI) was assessed using the 11-point Numeric Pain Rating Scale (NPRS), with 0 indicating No Pain and 10 indicating Worst Possible Pain. Approximately 1 hour before dosing and approximately 45 minutes before the 2-, 4-, and 6-hour time points, the participant rested for 45 minutes, then he or she started a treadmill walk at 15 minutes before dosing for baseline and at the 2-, 4-, and 6-hour time points, and then assessed ELEPI. Difference = predose (baseline) ELEPI score - ELEPI score 4 hours post dose.
Time Frame: Baseline, 4 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Part A) | Naproxen - 500 mg (Part A) | ADL5859 - 200 mg (Part A)
Number analyzed (Participants) | 45 | 45 | 45
units on a scale | 1.04 (1.437) | 1.72 (1.753) | 1.14 (1.553)

6. Secondary Outcome: Part A: Mean Peak Difference in ELEPI According to the NPRS Scale
Description: Evoked Lower Extremity Pain Intensity (ELEPI) was assessed using the 11-point NPRS. Participants were asked to rate their lower extremity pain on an 11 point NPRS, with 0 indicating No Pain and 10 indicating Worst Possible Pain. If a scheduled pain assessment was taken within 4 hours of rescue medication, the observed pain score was replaced by the pain score obtained right before the rescue medication was taken. Approximately 1 hour before dosing and approximately 45 minutes before the 2-, 4-, and 6-hour time points, the participant rested for 45 minutes, then he or she started a treadmill walk at 15 minutes before dosing for baseline and at the 2-, 4-, and 6-hour time points, and then assessed ELEPI. Peak ELEPID was defined as the maximum of ELEPIDs recorded at 2, 4, and 6 hours post dose. Difference = predose (baseline) NPRS score - peak NPRS score up to 6 hours post dose.
Time Frame: Baseline, Up to 6 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Part A) | Naproxen - 500 mg (Part A) | ADL5859 - 200 mg (Part A)
Number analyzed (Participants) | 45 | 45 | 44
units on a scale | 1.82 (1.874) | 2.49 (1.740) | 1.84 (1.725)

7. Secondary Outcome: Part A: Percentage of Participants in Each Treatment Group Achieving a 25%, 50%, or 75% Reduction From Baseline in Evoked Lower Extremity Pain Intensity Scores
Description: Percentage was measured by identifying the number of participants who achieved the desired percentage Reduction From Baseline in ELEPI Score at either 2, 4, and 6 hours post dose and was divided the by the number of total participants in the given group and then multiplied by 100 to equate to a percentage.
Time Frame: Up to 2, 4, and 6 hours post dosing
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo (Part A) | Naproxen - 500 mg (Part A) | ADL5859 - 200 mg (Part A)
Number analyzed (Participants) | 45 | 45 | 44
Percentage of Participants
  2 Hours Post-Dose, 25% Reduction | 28.9 | 46.7 | 22.7
  4 Hours Post-Dose, 25% Reduction | 40.0 | 60.0 | 36.4
  6 Hours Post-Dose, 25% Reduction | 42.2 | 64.4 | 45.5
  2 Hours Post-Dose, 50% Reduction | 4.4 | 24.4 | 4.5
  4 Hours Post-Dose, 50% Reduction | 22.2 | 31.1 | 15.9
  6 Hours Post-Dose, 50% Reduction | 26.7 | 33.3 | 18.2
  2 Hours Post-Dose, 75% Reduction | 0 | 6.7 | 0
  4 Hours Post-Dose, 75% Reduction | 0 | 8.9 | 6.8
  6 Hours Post-Dose, 75% Reduction | 6.7 | 11.1 | 6.8

8. Secondary Outcome: Part B: Participants' Global Evaluation of Study Medication
Description: For Part B, each participant's global evaluation (overall impression) of study medication was obtained at each weekly visit. Scores were recorded on the Case Report Form (CRF) on a 5 point scale ranging from "excellent" to "poor". Participant counts per score were reported at Week 1 (Day 7) and Week 2 (Day 14).
Time Frame: Up to Week 1 and Week 2
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Placebo (Part B) | ADL5859 - 100 mg (Part B)
Number analyzed (Participants) | 24 | 20
Participants
  Week 1 - Excellent (n=23, 20) | 2 | 3
  Week 1 - Very good (n=23, 20) | 5 | 7
  Week 1 - Good (n=23, 20) | 6 | 4
  Week 1 - Fair (n=23, 20) | 6 | 4
  Week 1 - Poor (n=23, 20) | 4 | 2
  Week 2 - Excellent (n=24, 19) | 2 | 4
  Week 2 - Very Good (n=24, 19) | 5 | 4
  Week 2 - Good (n=24, 19) | 7 | 3
  Week 2 - Fair (n=24, 19) | 5 | 5
  Week 2 - Poor (n=24, 19) | 5 | 3

9. Secondary Outcome: Part B: Mean Daily Average LEPI Scores Over the Last 24 Hours at Week 1 and Week 2
Description: Each day during Part B, participants rated their Lower Extremity Pain Intensity over the last 24 hours on an 11-point NPRS, with 0 indicating No Pain and 10 indicating Worst Possible Pain
Time Frame: Week 1 and Week 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Part B) | ADL5859 - 100 mg (Part B)
Number analyzed (Participants) | 24 | 20
units on a scale
  Week 1 | 4.66 (1.872) | 4.26 (1.741)
  Week 2 | 4.57 (2.197) | 4.25 (1.777)

10. Secondary Outcome: Part B: Mean Daily Average Overall Pain Intensity Scores Over Week 1, Over Week 2, and Over a 2-Week Period
Description: During Part B, participants returned to the clinic for 2 additional visits at approximately weekly intervals for assessments of Overall Pain Index (OPI). Participants rated their OPI on an 11-point Numeric Pain Rating Scale (NPRS) with 0 indicating No Pain and 10 indicating Worst possible pain
Time Frame: Baseline through Week 1, Week 1 through Week 2, and Baseline through Week 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Part B) | ADL5859 - 100 mg (Part B)
Number analyzed (Participants) | 24 | 20
units on a scale
  Change from Baseline to Week 1 | 4.26 (2.050) | 4.26 (1.939)
  Change from Week 1 to Week 2 | 4.33 (2.426) | 4.06 (1.955)
  Change from Baseline to Week 2 | 4.33 (2.125) | 4.21 (1.805)

11. Secondary Outcome: Part B: Percentage of Participants Using Rescue Medication
Description: The percentage of participants who took at least 1 dose of rescue medication during 2-week treatment period of Part B is presented.
Time Frame: Baseline through Week 2
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo (Part B) | ADL5859 - 100 mg (Part B)
Number analyzed (Participants) | 24 | 20
Percentage of Participants | 45.8 | 40.0

12. Secondary Outcome: Part A: Participant's Global Evaluation of Study Medication
Description: For each treatment period during Part A, each participant's global evaluation (overall impression) of study medication was obtained 6 hours after dosing. Scores were recorded on the Case Report Form (CRF) on a 5 point scale ranging from "excellent" to "poor". Participant counts per score were reported once in Part A.
Time Frame: 6 hours post dose during Treatment Periods 1, 2, and 3 of Part A
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo (Part A) | Naproxen - 500 mg (Part A) | ADL5859 - 200 mg (Part A)
Number analyzed (Participants) | 45 | 45 | 44
participants
  Excellent | 1 | 6 | 1
  Very Good | 9 | 12 | 8
  Good | 15 | 15 | 12
  Fair | 12 | 9 | 15
  Poor | 8 | 3 | 8

13. Primary Outcome: Part B: The Mean of Daily Average "Now" Lower Extremity Pain Intensity (LEPI) Score During the 2-Week Period
Description: Participants assessed their "Now" LEPI 3 times each day (morning, midday, and evening at approximately 10 AM, 2 PM, and 8 PM) and before taking any rescue medication. At each time point, participants were asked to rate their lower extremity pain on an 11-point Numeric Pain Rating Scale (NPRS), with 0 indicating No Pain and 10 indicating Worst Possible Pain. If a scheduled pain assessment was taken within 4 hours of rescue medication, the observed pain score was replaced by the pain score obtained right before the rescue medication was taken.
  LS means and SE were calculated from an analysis-of-covariance model with effect for treatment and baseline "Now" LEPI (before dosing for Treatment Period 1 of Part A) as a covariate. Participants with no postbaseline assessments were excluded from the baseline summary.
Time Frame: Baseline through 2 Weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Part B) | ADL5859 - 100 mg (Part B)
Number analyzed (Participants) | 24 | 20
units on a scale | 4.23 (0.339) | 4.21 (0.371)

ADVERSE EVENTS:
Description: Analysis Population:
  All participants who received at least 1 dose of study drug
Arm/Group | Placebo (Part A) | Naproxen - 500 mg (Part A) | ADL5859 - 200 mg (Part A) | Placebo (Part B) | ADL5859 - 100 mg (Part B)
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46 | 0/46 | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 8/46 | 7/46 | 8/46 | 10/24 | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A) (N=46) | Naproxen - 500 mg (Part A) (N=46) | ADL5859 - 200 mg (Part A) (N=46) | Placebo (Part B) (N=24) | ADL5859 - 100 mg (Part B) (N=20)
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 1 | 1 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Heart Rate Increase (Investigations) | 0 | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 2 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Abnormal Dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 2 | 2 | 3 | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Chest Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza-like Disorder (General disorders) | 0 | 0 | 0 | 0 | 1
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Haematocrit Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Red Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other